CLINICAL TRIAL: NCT00930410
Title: Intra-ductal Confocal Endomicroscopy for Characterization of Pancreas and Bile Duct Tumor
Acronym: EMID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EMID/IPC 2008-001
Record Dates: First submitted 2009-06-27; First posted 2009-06-30 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Pancreas Neoplasms; Bile Duct Diseases
Keywords: pancreas neoplasms; bile duct diseases; Cholangiopancreatography, Endoscopic Retrograde; ERCP
MeSH Terms: conditions — Pancreatic Neoplasms; Bile Duct Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- endomicroscopy (Experimental): Utilisation of an intra-ductal confocal endomicroscopy during the endoscopic Retrograde Cholangio-Pancreatography
  Interventions: Procedure: Endoscopic Retrograde Cholangio-Pancreatography (ERCP)

INTERVENTIONS:
Procedure: Endoscopic Retrograde Cholangio-Pancreatography (ERCP) — Utilisation of the Intra-ductal confocal endomicroscopy to obtain any exploitable image for the anatomopathology.

SUMMARY:
The endomicroscopy is an adaptation of traditional optical microscopy in the digestive endoscopy. Furthermore, with the integration of a miniaturized laser confocal microscope to a videoendoscope, it's possible to study the digestive mucous by "optical biopsy". This monocentric, non randomized and prospective study uses the Intra-ductal confocal endomicroscopy for the characterization of pancreas and bile duct tumor.

DETAILED DESCRIPTION:
Primary objective:

Obtain a tissular characterization of a biliary or pancreatic stenosis with a confocal microscope which is in direct contact of the stenosis during the Endoscopic Retrograde Cholangio-Pancreatography (ERCP).

Secondary objectives:

* Compare the result of this "optical biopsy" to a conventional biopsy.
* Tolerance

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to older
* Patient with an inflammatory or tumoral stenosis of bile duct or a solid or cystic tumor in the pancreas with a dilatation of the principal pancreatic canal.
* Signed consent

Non inclusion Criteria:

* Patient who have no indication for an ERCP
* Allergy to fluorescein
* Allergic rhinitis, asthma, eczema
* Pregnancy, breast feeding
* Patients with dialysis
* Patient with severe heart failure
* Patient with cirrhosis
* Hemostasis failure which can induce difficulties or contraindication for the biopsy during the conventional endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The principal outcome is the percentage of successful in vivo examination according to the localisation of the stenosis. A successful examination is defined by the obtention of exploitable image for the anatomopathology. | 2 days

SECONDARY OUTCOMES:
Study of the concordance between optical and histological biopsy | 2 days
Frequency and grade of adverse effects induced by the confocal endomicroscopy | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Marc GIOVANNINI, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (2):
- Institut PAOLI-CALMETTES, Marseille, France
- Centre Hospitalier Princesse Grasse, Monaco, Monaco

REFERENCES:
- See also: Official web site of the sponsor — http://www.institutpaolicalmettes.fr/